CLINICAL TRIAL: NCT04832529
Title: A Perianal Abscess Cavity Packing Versus no Packing; a Randomized Control Trial.
Brief Title: A Perianal Abscess Cavity Packing vs no Packing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Lajpat Rai, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-1537/DUHS/Approval/2020
Record Dates: First submitted 2021-03-21; First posted 2021-04-05 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Perianal Abscess; Ischiorectal Abscess

STUDY DESIGN:
Intervention Model Description: Experimental Randomized Control Trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perianal abscess cavity packing (Active Comparator)
  Interventions: Procedure: No packing of perianal abscess cavity
- Perianal abscess cavity no packing (Experimental)
  Interventions: Procedure: No packing of perianal abscess cavity

INTERVENTIONS:
Procedure: No packing of perianal abscess cavity — introducing new method to no packing of abscess cavity.

SUMMARY:
This prospective randomized trial will be conducted in all patients undergoing packing or no packing for perianal abscess cavity after incision and drainage, for 6 months after approval from IRB in Surgical unit III, Civil Hospital Karachi. Patient will be selected simple random sampling technique based on inclusion criteria. Patient will be assessed for post-operative pain, healing of cavity and recurrence of abscess. At first time of debridement pus or tissue will be sent for culture and sensitivity, meanwhile broad-spectrum antibiotic will be started.

Questionnaire will be filled by PI for post-operative pain, recurrence of abscess, quality of life, wound healing, post operative fistula in ano and chronic post surgical pain either due to packing or no packing.

DETAILED DESCRIPTION:
This is an experimental randomized control trial will start 6 months after approval from Institution Review Board. All patients with perianal abscess after incision and drainage cavity will be either packed or not after informed consent. Pack will be changed daily as regular dressing till healing occurs. Packing reduces bleeding and heals cavity by effect of dressing solution in which gauze is soaked. Other group with dressing will be changed daily and will be assessed for healing week. There is no pain in simple dressing applied over cavity. Patient will receive broad spectrum antibiotics according to pus or tissue culture. During this period, laboratory investigation CBC, CRP will be sent to check the response. Sits bath will be advised to both groups. Post-operative pain, cavity healing will be assessed by faculty.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Age less than 70 years
* Perianal abscess

Exclusion Criteria:

* Suspected inflammatory bowel disease
* Fournier's gangrene
* Horseshoe/bilateral abscess

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 14 days
  Pain will be assessed via visual analogue scale from 1-10 while changing of dressing.

SECONDARY OUTCOMES:
Decreases hospital visit | 3 weeks
  Hospital visits will be decreased when dressing only dressing to be done, not wound packing.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Ruth K.M Pfau Civil Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No